CLINICAL TRIAL: NCT02029677
Title: Putative Hormonal Mechanisms of Appetite Suppression Following LAGB: A Pilot Study
Brief Title: Appetite Suppression / Hormone Study Control Group
Status: Active, not recruiting | Type: Observational
Sponsor: Oregon Weight Loss Surgery, LLC (Other)
Collaborators: Legacy Health System (Other); Allergan (Industry)
Responsible Party: Principal Investigator, Emma Patterson, Emma Patterson, M.D., Oregon Weight Loss Surgery, LLC
Other Study IDs: FWA00001280
Record Dates: First submitted 2013-12-18; First posted 2014-01-08 (Estimated); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Morbid Obesity; Bariatric Surgery Patient
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Each time these hormone assays are performed, aliquots of plasma will be frozen at -80C:
  * Total immunoreactive ghrelin - Plasma will be assayed in duplicate for immunoreactive ghrelin concentration using a commercial radioimmunoassay (RIA)
  * Lipids - Plasma total cholesterol, TG, HDL-C, and LDL-C will be measured
  * Glucose and insulin - Plasma glucose concentrations will be measured in triplicate using the glucose oxidase method. Plasma insulin will be measured in duplicate using a modification of a double antibody radioimmunoassay
  * Adiponectin and other gut hormones - Adiponectin, PYY3,36 and GLP-1 will be measured using a commercial RIA. Pancreatic polypeptide (PP) will be measured using a commercial RIA
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to determine how changes in levels of obesity-related hormones in the gastrointestinal tract following Laparoscopic Adjustable Gastric Banding (LAGB) surgery may lead to a decrease in appetite and weight loss. Learning exactly how the Lap Band works may help us to develop new, less invasive treatments for morbid obesity. This knowledge may also lead to the development of preventive, cost-effective treatment strategies. As a control subject, participants will provide a comparison for changes in these hormones with medical weight loss compared to weight loss after LAGB surgery.

DETAILED DESCRIPTION:
The expected duration of participation in the study is up to 6 months before bariatric surgery depending on participants' weight loss and insurance company requirements. A total of 10 patients will take part in this control group.

The following procedures and tests will be done before surgery: routine standard tests required to be involved in the obesity surgery program (history and physical, blood work, ECG, nutritional assessment, psychological assessment and sleep study). During preoperative evaluation participants will be started on a medical weight loss diet with instructions provided by the program's endocrinologist, nurse practitioners and dietitians with the weight loss goals as stipulated by insurance companies and have a series of additional laboratory tests (blood work) done to test the hormonal response to weight loss.

This blood work, which is drawn after eating a standardized meal, is the only experimental procedure of the entire study. We will be measuring several hormones associated with obesity including ghrelin, obestatin, peptide tyrosine tyrosine (PYY3-36), adiponectin, Glucagon-like peptide-1 (GLP-1), oxyntomodulin, leptin, insulin, glucose and pancreatic polypeptide (PP). Measurements will be done at 4 time intervals before surgery: at enrollment, +1-month, +3-months, and +6-months. This will allow us to look at hormone levels as participants gradually lose weight. If a participant reaches the insurance-dictated weight loss before 6 months, study participation will cease to allow the individual to proceed with surgery scheduling.

Participants will be required to fast overnight prior to each visit. An intravenous line will be placed at 0800, all subjects will be fed a standard breakfast (35% fat, 15% protein, and 50% carbohydrate) consisting of 25% of estimated caloric needs for weight maintenance, which they will consume in 30 minutes or less. Blood will be taken beginning 30 minutes before the standardized meal, then at time 0, then 30, 60, 90, and 120 minutes after the meal for total ghrelin, pancreatic polypeptide, PYY3-36, active GLP-1, insulin, glucagon, leptin, oxyntomodulin, and glucose. An extra fasting sample will be obtained for lipids and total adiponectin. Three-quarters of a cup (148 mL) of blood will be drawn for analysis at each visit. Additionally, subjects will be asked to complete a Visual Analog Scale (VAS) three times during each research visit by placing a single vertical mark across a 100 mm in length line, with words anchored at each end, expressing the most positive and the most negative rating, to assess hunger, satiety, and fullness. Each visit will last approximately 4 hours.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of equal to or greater than 35 kg/m2, and less than 60 kg/m2
* Age great than or equal to 18 years and less than 70 years
* Able to provide informed consent
* If female with reproductive potential, agrees to use a reliable method of birth control for the duration of the study (6 months)

Exclusion Criteria:

* Enrolled in another clinical study which involves an investigational drug
* Any condition where protocol compliance is unlikely (e.g. anxiety disorder, inadequate comprehension)
* Pregnancy
* Previous gastric or esophageal surgery
* Immunosuppressive drugs including corticosteroids
* Type 2 diabetes
* Coagulopathy (INR > 1.5 or platelets < 100,00/ul)
* Anemia (Hgh < 10.0 g/dl)
* Any contraindication to treatment
* A severe concurrent illness likely to limit life (e.g. cancer)
* Significant malabsorptive or gastrointestinal disorder (e.g. pancreatic insufficiency, Celiac sprue, or Crohn's disease)

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with morbid obesity or severe obesity with comorbidities who meet the National Institutes of Health criteria for bariatric surgery and required by insurance to participate in a medically supervised weight loss program prior to authorization for surgery will be offered enrollment into the study. The 10 subjects enrolled will be men and women ages 18 to 69 years with a BMI of greater than or equal to 35 kg/m2 and less than 60 kg/m2. Patients must be fit to undergo major abdominal surgery and be reasonably expected to complete the six-month study protocol prior to authorization for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2008-09; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Hormonal Mechanism of Action for Weight Loss | Preoperatively (baseline) and at 1-, 3- and 6-months post-surgery
  Our primary outcome measures the mechanism of action of the adjustable band in producing weight loss from the time of surgery to visit timepoints at plus one, 3 and six months following LAGB placement. Changes in appetite and hunger will be measured in the form of a validated clinical analogue scale from baseline to 1, 3 and 6 months post-surgery. Statistical analysis will be performed to look for changes in blood levels of gut hormones (total ghrelin, PYY3-36, total adiponectin, active GLP-1, glucose, glucagon, insulin, leptin, oxyntomodulin, and pancreatic polypeptide) measured before and after a standardized meal from baseline values to 1, 3, and 6 months post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Emma J Patterson, MD, Principal Investigator — Oregon Weight Loss Surgery
Locations (1):
- Oregon Weight Loss Surgery, Portland, Oregon, United States